CLINICAL TRIAL: NCT00968630
Title: Human Immunodeficiency Virus (HIV)-Specific Immune Reconstitution After Hematopoietic Cell Transplant for Treatment of Hematologic Malignancy in Patients Infected With HIV
Brief Title: Immune Response After Stem Cell Transplant in HIV-Positive Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2212.00; NCI-2009-01244 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2212; 2212.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA018029 (NIH); P30CA015704 (NIH); U19AI096111 (NIH)
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; HIV Infection
MeSH Terms: conditions — Hematologic Neoplasms; HIV Infections | interventions — Leukapheresis

ARMS (1):
- Treatment (HIV-specific immune reconstitution after HCT) (Experimental): Patients undergo leukapheresis for analysis of HIV-1 latent reservoir at baseline and at days +90, +180, +365, and +730, and then annually thereafter as feasible.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Leukapheresis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis

SUMMARY:
This phase II trial studies the immune response after stem cell transplant in human immunodeficiency virus (HIV)-positive patients with hematologic cancer (blood cancer). Studying samples of blood from HIV-positive patients with cancer in the laboratory may help doctors learn more about changes that occur in the immune system after stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the development of donor-derived HIV-1-specific immune response following hematopoietic cell transplant (HCT) for treatment of hematologic malignancy in HIV+ patients.

II. Examine the affect of HCT on the pool of latently infected cluster of differentiation (CD)4+ T cells in HIV+ patients given HCT for treatment of hematologic malignancy.

OUTLINE:

Patients undergo leukapheresis for analysis of HIV-1 latent reservoir at baseline and at days +90, +180, +365, and +730, and then annually thereafter as feasible.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Treatment with highly active antiretroviral therapy (HAART) for at least 1 month
* Viral load has decreased by >= 1.5 logs or viral load < 5000 copies/ml plasma on HAART therapy
* Hematologic malignancy associated with a poor prognosis or other diagnosis for which hematopoietic cell therapy (allogeneic or autologous, including gene therapy) is indicated
* Approval for allogenic regimen given at Patient Care Conference
* DONOR: Autologous or allogeneic gene modified cells allowed

Exclusion Criteria:

* A medical history of noncompliance with HAART or medical therapy
* Inability to provide informed consent
* DONOR: Allogeneic donors must not have HIV infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-12-17 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
Quantification of donor-derived HIV-1-specific immune responses following HCT | Up to 1 year
  HIV-1 specific immune responses will be evaluated in samples collected before and after HCT. These results will be used descriptively.
Quantification of latently infected CD4+ cells in HIV+ patients | Up to 7 years
  The overall measure of efficacy will be the log change in HIV-1 latent reservoir, measured as infectious units per million.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Woolfrey, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States